CLINICAL TRIAL: NCT04553900
Title: Effect of Heat Stress on Global LV Function in Anesthetized Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Edward O'Brien, Associate Professor of Anesthesiology, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 171159
Record Dates: First submitted 2020-09-11; First posted 2020-09-18 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Hyperthermia; Cardiac Functional Disturbances During Surgery
MeSH Terms: conditions — Hyperthermia | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transesophageal Echocardiography — Placement of a transesophageal probe and performance of a diagnostic Transesophageal echocardiography examination.

SUMMARY:
Recent data suggests that increased temperature improves inotropic function during systole and may improve diastolic function in healthy humans at rest, despite a reduction in left ventricular volume at end diastole. The effect of heat stress has not been reported in patients receiving general anesthesia and the impact of general anesthesia on these findings is not known. Trans-esophageal echocardiography will be used to measure parameters important to both systolic and diastolic function at temperature intervals of 1°C in patients undergoing "Heated Intraoperative Peritoneal Chemotherapy" (HIPEC.) That general anesthesia will not alter the cardiovascular effects of increased temperature that has been reported in healthy, un-anesthetized humans is the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* any patient presenting for hyperthermic intraperitoneal chemotherapy.

Exclusion Criteria:

* Subjects less than 18 years old.
* pregnant women
* prisoners,
* institutionalized individuals
* Any patient with known contraindication to Transesophageal echocardiography.
* Patients with known cardiac dysfunction prior to screening will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Change in ejection fraction before and after hyperthermia | Approximately 6 hours from prior to hyperthermia to during hyperthermia.

SECONDARY OUTCOMES:
Transmitral inflow velocities before and after hyperthermia | Approximately 6 hours from prior to hyperthermia to during hyperthermia.
Pulmonary venous inflow velocities before and during hyperthermia | Approximately 6 hours from prior to hyperthermia to during hyperthermia.
Mitral annular tissue doppler velocities before and during hyperthermia | Approximately 6 hours from prior to hyperthermia to during hyperthermia.

OTHER OUTCOMES:
heart rate before and during hyperthermia | Approximately 6 hours from prior to hyperthermia to during hyperthermia.
mean arterial pressure before and during hyperthermia | Approximately 6 hours from prior to hyperthermia to during hyperthermia.

CONTACTS AND LOCATIONS:
Overall Officials: Edward O O'Brien, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No